CLINICAL TRIAL: NCT01921231
Title: Selective Subarachnoid Anesthesia. Comparison of Hyperbaric Bupivacaine and Hyperbaric Prilocaine in Knee Arthroscopy and Inguinal Hernia Repair in Ambulatory Surgery
Brief Title: Selective Subarachnoid Anesthesia. Comparison of Hyperbaric Bupivacaine and Hyperbaric Prilocaine
Acronym: BUPIPRILO-07
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Pere Roura-Poch (Other)
Responsible Party: Sponsor-Investigator, Dr. Pere Roura-Poch, Head of Clinical epidemiology department, Consorci Hospitalari de Vic
Organization: Consorci Hospitalari de Vic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-006930-17
Record Dates: First submitted 2013-08-01; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Knee Arthroscopy (for Diagnostic or Therapy); Inguinal Hernia Repair (Not Urgent)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric prilocaine 1% (Experimental): Solution for injection. Intradural use. In order to obtain Prilocaine 1% we charge a syringe with 2 mL Prilocaine 2%, and we add 1 mL Saline solution (0.9%) and 1 mL Glucose solution (33%). Administer 3 mL of syringe contains in two minutes.
  Interventions: Drug: Hyperbaric Prilocaine 1%
- Hyperbaric Bupivacaine 0.5% (Active Comparator): Solution for injection. Intradural use. Charge a syringe with 1 mL of Bupivacaine (0.5%) and administer it in a minute.
  Interventions: Drug: Hyperbaric bupivacaine 0.5%

INTERVENTIONS:
Drug: Hyperbaric Prilocaine 1% — Selective spinal anesthesia was performed on induction-block area and patient was transferred to the assigned operating room where another anesthesiologist (blinded for the arm) began to evaluate the blocking. Neither the nurse, surgeon nor the anesthesiologist involved in the patient evaluation knew the allocation group.
  Arms: Hyperbaric prilocaine 1%
Drug: Hyperbaric bupivacaine 0.5% — Selective spinal anesthesia was performed on induction-block area and patient was transferred to the assigned operating room where another anesthesiologist (blinded for the arm) began to evaluate the blocking. Neither the nurse, surgeon nor the anesthesiologist involved in the patient evaluation knew the allocation group.
  Arms: Hyperbaric Bupivacaine 0.5%

SUMMARY:
Selective spinal anesthesia is widely used for ambulatory surgery. Unilateral spinal anesthesia is a suitable option for ambulatory anesthesia as it is efficient and effective. Lidocaine has been the well-known choice for this procedure. However, it is associated to transient neurologic symptoms (TNS). Different anesthetic strategies for this procedure have been performed, for example, the use of small doses of long-acting agents and the use of additives such as opioids. The ideal local anesthetic should be lidocaine-like without risk of transient neurologic symptoms. We design and plan a randomised clinical trial to show if hyperbaric prilocaine 2% would be an alternative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a scheduled knee arthroscopy
* Patients with a scheduled inguinal hernioplasty

Exclusion Criteria:

* Patient refusal to regional anesthesia
* American Society of Anesthesiologists score risk equal or greater than 4
* Body mass index greater than 32
* Coagulopathy
* Cutaneous infection at injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-05; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Length of stay in post-operative care unit (in minutes) | Participants will be followed an average of 6 hours from surgical incision closure to accomplish discharge criteria to go home
  Time in minutes from closing the surgical incision until to having criteria for discharge to home.

SECONDARY OUTCOMES:
Level of motor blocking | At surgical incision and at 60 minutes after anesthesia
  Assessed by Bromage score who ranges from Complete block (unable to move feet or knees, score 1) to Able to perform partial knee bend (score 6 who means nil block).
Fast-track (by-pass recovery area) | Participants will be assessed when surgical incision is closed with surgical staples
  Number (and percentage) of patients in each arm that can be transferred directly from the operating room to postsurgical ward. A minimal score of 12 (on modified Aldrete's scoring system with no score <1 in any individual category) would be required for a patient to be fast-tracked.
Peak sensory block level | One minute before surgical incision
  The sensory block level was determined pricking dermatomes with a pin from down to up.
Transient neurological symptoms | At hospital discharge (an average of 8 hours after admission), and at home at 24, 48 and 72 hours after surgery
  Researchers surveyed if appears pain originated in gluteal region and radiating to both lower extremities following patients by phone.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Serrat-Puyol, MD, Study Director — Vic Hospital Consortium; Pere Roura-Poch, MD, MPH, Study Chair — Vic Hospital Consortium
Locations (1):
- Vic Hospital Consortium, Vic, Catalonia, Spain